CLINICAL TRIAL: NCT02379273
Title: The Nucleus Hybrid L24 Implant System: Extended Duration Post Approval Study
Brief Title: Nucleus Hybrid L24 Extended Duration Post Approval Study
Acronym: HED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: University of Iowa (Other); NYU Langone Health (Other); Midwest Ear Institute (Other); University of Cincinnati (Other); The Center for Hearing and Balance Disorders (Ambiguous); Ohio State University (Other); Mayo Clinic (Other); Hearts for Hearing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-5563-HYB-PMA
Record Dates: First submitted 2015-01-29; First posted 2015-03-04 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hybrid L24 pivotal study subjects (Experimental): Subjects implanted with the Nucleus Hybrid L24 Implant as part of the pivotal IDE study and who still have the device implanted will continue to be followed for 5 years post activation
  Interventions: Device: Nucleus Hybrid L24 Implant

INTERVENTIONS:
Device: Nucleus Hybrid L24 Implant — Subjects have already been implanted with the Nucleus Hybrid L24 implant.

SUMMARY:
This post approval study evaluates the long term safety and efficacy of the Nucleus Hybrid L24 Implant System in a group of already implanted recipients.

DETAILED DESCRIPTION:
The Hybrid L24 Implant System (P130016) was the subject of a pivotal clinical trial (IDE G070191) from 2007 through 2012. Data on the 50 subjects enrolled in the study, in support of safety and efficacy of the device, was submitted in June 2013 as part of Premarket Approval (PMA) #130016. As a condition of approval, March 20, 2014, a Post-Approval Study was designed to monitor the long-term (5 years postactivation for each subject) safety and effectiveness of the device in this existing cohort of implanted subjects was designed.

ELIGIBILITY:
Inclusion Criteria:

- Recipients who were implanted with the Hybrid L24 as part of the original pivotal IDE study

Exclusion Criteria:

* Recipients who withdrew or were terminated from the L24 pivotal IDE study
* Recipients who were re-implanted and no longer have a Nucleus Hybrid L24 implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Gantz, MD, Principal Investigator — University of Iowa

REFERENCES:
- [Derived] Reinhart PN, Parkinson AJ, Dunn CC, Gantz BJ. Factors Affecting Audiometric and Speech Perception Outcomes in Hybrid Cochlear Implant Recipients. Laryngoscope. 2025 Oct 8. doi: 10.1002/lary.70195. Online ahead of print. PMID 41059917
- [Derived] Roland JT Jr, Gantz BJ, Waltzman SB, Parkinson AJ. Long-term outcomes of cochlear implantation in patients with high-frequency hearing loss. Laryngoscope. 2018 Aug;128(8):1939-1945. doi: 10.1002/lary.27073. Epub 2018 Jan 13. PMID 29330858

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight of 10 pivotal study sites agreed to participate.
  All subjects who remained enrolled under the pivotal Investigational Device Exemption (IDE) study (G070191) or under a continued access study (G070191/S024) were eligible to participate in this post-approval study.
  Subject enrollment for this study was completed in the period, January 14, 2015 through September 12, 2016.
Pre-assignment Details: Of 53 subjects implanted prior to this study: 6 no longer used the Hybrid L24 implant, 8 subjects were not available to enroll, and 4 subjects declined participation.
  Thirty-five subjects enrolled in this postapproval study. First subject enrolled January 14, 2015; last subject enrolled September 12, 2016.
Groups:
- Hybrid L24 Pivotal Study Subjects.: Available subjects implanted under the pivotal IDE study (G070191) or under a continued access study (G070191/S024) were followed for 5 years postactivation.
Period: Overall Study
Arm/Group | Hybrid L24 Pivotal Study Subjects.
Started | 35
Completed | 35 (Completed 5 years postactivation.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hybrid L24 Pivotal Study Subjects.
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35
Aided Speech Recognition [Mean (Standard Deviation); unit: Percentage of total words correctly re] — Aided speech perception refers to the percentage of total words correctly recognized for the speech material presented from a loudspeaker, with the subjects using amplification (i.e., hearing aids).
  Percentage of total words correctly re
    CNC Words Implanted Ear: Percentage of total words correctly recognized. | 27 (14.6)
    CNC Words Bilateral: Percentage of total words correctly recognized. | 44.4 (17.3)
    CNC Words Contralateral: Percentage of total words correctly recognized. | 39 (17.9)
    AzBio+5 dB SNR Implant Ear: Percentage of total words correctly recognized. | 15.7 (13.7)
    AzBio+5 dB SNR Bilateral: Percentage of total words correctly recognized. | 28.8 (20.6)

OUTCOME MEASURES:

1. Primary Outcome: Consonant-Nucleus-Consonant (CNC) Word Recognition in Quiet: Percentage of Total Words Correctly Recognized.
Description: The CNC Words test consists of 10 recorded lists of 50 monosyllabic words in compact disk format. For this study, two lists were administered in quiet at a level equal to 60 dBA (decibels A-weighted) in the sound field and scored as total number of words correct, which will be expressed as a percentage correct. Minimum score is 0/100 words or 0% (worse), maximum score is 100/100 or 100% (best possible).
Time Frame: 5 years postactivation.
Population: All subjects completing the 5-year postactivation evaluation interval.
Measure: Mean (Standard Deviation); unit: percentage of total words correct
Arm/Group | Hybrid L24 Pivotal Study Subjects.
Number analyzed (Participants) | 35
percentage of total words correct
  Implanted Ear | 71.2 (20.4)
  Bilateral Condition | 81 (12.7)
Statistical Analysis 1: Comparison: Hybrid L24 Pivotal Study Subjects; A Friedman repeated-measures ANOVA on ranks was applied to the unilateral CNC data with follow-up pairwise comparisons based on the Tukey Test; Test type: Superiority; p < 0.001, ANOVA — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Hybrid L24 Pivotal Study Subjects; Test type: Superiority — A Friedman repeated-measures ANOVA on ranks was applied to the bilateral CNC data with follow-up pairwise comparisons based on the Tukey Test; p < 0.001, ANOVA — The threshold for statistical significance was p = 0.05

2. Primary Outcome: AzBio (Arizona Biomedical Institute) Sentence Recognition in Noise: Percentage of Total Words Correctly Recognized.
Description: The AzBio Sentence Test consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in' unintelligible words. Each list includes 5 sentences from 4 different male and female speakers. Each word in the sentence counts towards the overall score. Minimum score is 0 out the total number of words in a given list (varies list to list, with an average length of 141 words) words or 0% (worse), maximum score is all words correctly repeated or 100% (best possible).
Time Frame: 5 years postactivation.
Population: All subjects completing the 5-year postactivation evaluation interval.
Measure: Mean (Standard Deviation); unit: percentage of total words correct
Arm/Group | Hybrid L24 Pivotal Study Subjects.
Number analyzed (Participants) | 35
percentage of total words correct
  Implanted Ear | 49.6 (27.5)
  Bilateral Condition | 61.4 (24.5)
Statistical Analysis 1: Comparison: Hybrid L24 Pivotal Study Subjects; Test type: Superiority — A Friedman repeated-measures ANOVA on ranks was applied to the unilateral AzBio data with follow-up pairwise comparisons based on the Tukey Test; p < 0.001, ANOVA — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Hybrid L24 Pivotal Study Subjects; Test type: Superiority — A Friedman repeated-measures ANOVA on ranks was applied to the bilateral AzBio data with follow-up pairwise comparisons based on the Tukey Test; p < 0.001, ANOVA — The threshold for statistical significance was p = 0.05

3. Post Hoc Outcome: Speech, Spatial and Qualities of Hearing Scale (SSQ): Speech Hearing Subscale
Description: The Speech, Spatial, and Qualities of Hearing Scale or SSQ (Gatehouse & Noble, 2004) was administered as a self-assessment of hearing (dis)abilities across a range of listening situations that fall within three hearing domains: Speech Hearing, Spatial Hearing, and Qualities of Hearing.
  Within each domain or subscale, each question is scored by the reader indicating on a line marked from 0 through 10. The score for each subscale represents the average of the responses made to each question within the subscale. A score of zero is the minimum and corresponds to minimal ability (i.e., poorer) and 10 corresponds to complete ability (i.e., better) for each subscale.
Time Frame: Preoperative through 5 years postactivation.
Population: All subjects completing the 5-year postactivation evaluation interval.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid L24 Pivotal Study Subjects.
Number analyzed (Participants) | 35
score on a scale
  Preoperative | 3.3 (1.4)
  1 Year Postactivation | 5.9 (1.7)
  5 Years Postactivation | 5.4 (1.6)
Statistical Analysis 1: Comparison: Hybrid L24 Pivotal Study Subjects; Test type: Superiority — A one-way repeated-measures analysis of variance was applied to the data, with follow-up pairwise comparisons based on the Holm-Sidak method; p < 0.001, ANOVA — The threshold for statistical significance was p=0.05

4. Post Hoc Outcome: Speech, Spatial and Qualities of Hearing Scale: Spatial Hearing Subscale
Description: as for outcome 3
Time Frame: Preoperative through 5 years postactivation.
Population: All subjects completing the 5-year postactivation evaluation interval.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid L24 Pivotal Study Subjects.
Number analyzed (Participants) | 35
score on a scale
  Preoperative | 4.2 (1.8)
  1 Year Postactivation | 5.6 (2.0)
  5 Years Postactivation | 5.01 (1.7)
Statistical Analysis 1: Comparison: Hybrid L24 Pivotal Study Subjects; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.001, ANOVA; The threshold for statistical significance was p=0.05

5. Post Hoc Outcome: Speech, Spatial and Qualities of Hearing Scale: Qualities of Hearing Subscale
Description: as for outcome 3
Time Frame: Preoperative through 5 years postactivation.
Population: All subjects completing the 5-year postactivation evaluation interval.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid L24 Pivotal Study Subjects.
Number analyzed (Participants) | 35
score on a scale
  Preoperative | 4.8 (1.5)
  1 Year Postactivation | 6.7 (1.7)
  5 Years Postactivation | 6.4 (1.4)
Statistical Analysis 1: Comparison: Hybrid L24 Pivotal Study Subjects; Test type: Superiority — Pre- and postoperative mean scores were compared based on Friedman repeated-measures analysis of variance with follow-up pairwise comparisons based on the Tukey Test; p < 0.001, ANOVA — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were captured from baseline for this study through 5 years postactivation. Since subjects were recruited following their completion of the pivotal study baseline was anywhere from 2 years through 5 years postactivation.
Arm/Group | Hybrid L24 Pivotal Study Subjects.
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 3/35
Other Adverse Events (participants affected / at risk) | 4/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid L24 Pivotal Study Subjects. (N=35)
Heart Attack (Cardiac disorders) | 1 (1) — Subject reported to have had a heart attack prior to the 5-year postactivation evaluation. Subject was hospitalized to have stents placed, hence the adverse event (AE) was deemed serious. This AE was unrelated to the study device.
Cochlear implant revision (Ear and labyrinth disorders) | 1 (1) — Subject experienced a change in hearing and elected to have the Hybrid L replaced with a traditional cochlear implant 8 years after receiving the Hybrid implant.
Cochlear implant revision (Ear and labyrinth disorders) | 1 (1) — Subject had revision surgery to replace a contralateral Hybrid L implant, placed after Hybrid approval, associated with loss of residual hearing. Not related to the study device or procedure since it involved the non-study ear.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid L24 Pivotal Study Subjects. (N=35)
Teeth cracking and pain associated with Bruxism (General disorders) | 1 (1) — At study baseline, subject reported teeth cracking associated with pre-existing condition, bruxism (clenching of the teeth/jaw during sleep). Related to a pre-existing condition and not procedure/device related.
Ear pain (Ear and labyrinth disorders) | 1 (1) — Subject reported soreness under the external processor coil during a routine follow-up visit. Resolved with lower magnet setting.
Tinnitus (Ear and labyrinth disorders) | 1 (1) — After 6 years of device use, subject reported new low-frequency pulsatile tinnitus that occurred intermittently for a few hours daily in the implanted ear. Not device or procedure related as tinnitus present without device use.
Ear pain (Ear and labyrinth disorders) | 1 (1) — During final study visit, subject reported a sore and pain on top of pinna. Resolved with use of moleskin on ear hook.
Perceived change in hearing due to wax occlusion (Ear and labyrinth disorders) | 1 (1) — Wax occlusion resulting perceived decreased hearing in right (contralateral) ear, and feeling of water in ear. Resolved following removal of wax. Not related to study ear.

LIMITATIONS AND CAVEATS:
The non-study group presents a potential bias because it was comprised of a number who experienced significant changes in low-frequency acoustic hearing during the pivotal study and their outcomes beyond the pivotal study were not followed. Prior to the beginning of the post-approval study, 13 of the 18 subjects experienced profound/total loss of hearing between surgery and 18 months postactivation, compared with 9 of the 35 subjects who proceeded into the post-approval study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-09-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT02379273/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT02379273/SAP_001.pdf